CLINICAL TRIAL: NCT03729414
Title: Multicenter Randomized Controlled Trial of Doppler Guided Hemorrhoid Artery Ligation (DGHAL) and Mucopexy Versus Mucopexy Alone in the Treatment of Grade III Hemorrhoids
Brief Title: Doppler-guided or Non Doppler-guided Arterial Ligation and Mucopexy for Third Degree Hemorrhoids: That is the Question
Acronym: HAMLeT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: siccr
Record Dates: First submitted 2018-05-31; First posted 2018-11-02 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Hemorrhoids Prolapse
Keywords: Hemorrhoid; Doppler; Mucopexy
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Intervention Model Description: Prospective, multi-centre, parallel-arm randomized controlled equivalence trial. Eligible patients will be randomized to either mucopexy without Doppler guided artery ligation or mucopexy with doppler guided hemorroidal artery ligation.
Who Masked: Outcomes Assessor
Masking Description: long term outcome will be evaluated by a third observer unaware of the type of surgery performed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mucopexy with Doppler artery ligation (Active Comparator): Doppler guided hemorrhoidal artery ligation and mucopexy: Group of patients with III degree hemorrhoids treated by THD or AMI device is introduced into the anal canal. The terminal branches of the rectal artery are detected by the Doppler 2-3 cm above the dentate line. The tip of the instrument is tilted and arteries ligated with a figure-of-eight suture inserted using a special needle-holder. After the haemorrhoid artery ligation, the suture is continued with 3/5 sutures applied 5 mm apart, making sure that the last is at least 5 mm above the dentate line. The suture is then tied to create a hemorrhoidopexy. The procedure is repeated after all artery ligations (6 ligations
  Interventions: Procedure: mucopexy with Doppler artery ligation
- mucopexy without Doppler artery ligation (Experimental): Non Doppler guided hemorrhoidal artery ligation and mucopexy: A lubricating gel is applied to the tip of the THD or the AMI device and, with the patient in the lithotomy position, the proctoscope is introduced into the anal canal. the mucopexy will start at two o'clock and repeated at 4, 6 8, 10, 12, in clockwise direction
  Interventions: Procedure: mucopexy without Doppler artery ligation

INTERVENTIONS:
Procedure: mucopexy with Doppler artery ligation — Hemorrhoids will be treated by mucopexy with Doppler guided hemorrhoids arteries ligation performed in all quadrants
  Other Names: DGHAL
  Arms: mucopexy with Doppler artery ligation
Procedure: mucopexy without Doppler artery ligation — Hemorrhoids will be treated by mucopexy alone performed in all quadrants
  Other Names: NON-DGHAL
  Arms: mucopexy without Doppler artery ligation

SUMMARY:
Hemorrhoidal disease is one of the most common proctological disease affecting the general population from the mid-teens onward with considerable implications for the National Health Service (NHS) both from an economic point of view and from surgeon's workload.Improved understanding of the pathogenesis of hemorrhoids and of the complications associated with excisional hemorrhoidectomy led to the invention of newer surgical procedures, including Doppler guided hemorrhoidal artery ligation (DGHAL).

This technique was introduced in 1995 by Morinaga et al. and consists in the use of a proctoscope with a Doppler transducer that detect the arterial structures.

Since DGHAL does not involve tissue excision, it is expected to be associated with reduced postoperative pain if compared with hemorrhoidectomy.

In the last decade several devices (THD and AMI/ HAL-RAR - Hemorrhoidal Artery Ligation and Recto Anal Repair) have been developed in order to improve and facilitate the execution of the technique, making easier the procedure.

The hypothesis of the study is that a simple mucopexy procedure by suture-fixation of anal cushion without the aim of a Doppler device, could be as effective as DGHAL and mucopexy to manage prolapsing grade III hemorrhoids.

DETAILED DESCRIPTION:
Prospective, multi-centre, parallel-arm randomized controlled equivalence trial. Eligible patients will be randomized to either mucopexy without Doppler guided artery ligation or mucopexy with doppler guided hemorroidal artery ligation.

Primary aim of the Hamlet trial is to demonstrate that mucopexy without DGHAL for grade III haemorrhoids have equivalent recurrence rate at 1 year follow up of DGHAL with mucopexy procedure

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic grade III hemorrhoids according to Goligher
* No other source of anal bleeding than hemorrhoids
* Written informed consent

Exclusion Criteria:

* Any previous hemorrhoid surgery
* Participants expressing clear preference for one of the interventions
* Pregnancy
* Inability to understand the informed consent
* Oral anticoagulants of congenital defects of the coagulation
* Patients with immunodepression (i.e. HIV)
* Other proctological diseases (fissures, fistulas, condyloma, etc)
* IBD involving the anus ore the rectum

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
percentage of recurrences of hemorrhoidal prolapse | 1 year follow up
  Recurrence is defined as persistent or recurrent hemorrhoidal prolapse and graded according to Goligher in 4 degrees

CONTACTS AND LOCATIONS:
Overall Officials: Donato F Altomare, Principal Investigator — University of Bari
Locations (1):
- Dept of Emergency and Organ transplantation - University of Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ratto C, Campenni P, Papeo F, Donisi L, Litta F, Parello A. Transanal hemorrhoidal dearterialization (THD) for hemorrhoidal disease: a single-center study on 1000 consecutive cases and a review of the literature. Tech Coloproctol. 2017 Dec;21(12):953-962. doi: 10.1007/s10151-017-1726-5. Epub 2017 Nov 24. PMID 29170839
- [Result] Bursics A, Morvay K, Kupcsulik P, Flautner L. Comparison of early and 1-year follow-up results of conventional hemorrhoidectomy and hemorrhoid artery ligation: a randomized study. Int J Colorectal Dis. 2004 Mar;19(2):176-80. doi: 10.1007/s00384-003-0517-9. Epub 2003 Jul 5. PMID 12845454

DOCUMENTS (1):
  • Study Protocol (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03729414/Prot_000.pdf